CLINICAL TRIAL: NCT04192279
Title: Monitoring and Guidance of Early Lactate Clearance Rate in Patients With Sepsis
Brief Title: Early Lactate Clearance Rate in Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Second Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Fei Tong, Director, The Second Hospital of Hebei Medical University
Other Study IDs: 78247891400
Record Dates: First submitted 2019-12-04; First posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Early Lactate Clearance
Keywords: sepsis; lactate; early
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- lactate group: Lactate early guide resuscitation
  Interventions: Diagnostic Test: lactate clearance
- control group: early guide resuscitation without lactate

INTERVENTIONS:
Diagnostic Test: lactate clearance — Lactate clearance rate was monitored within 6 hours after admission
  Groups: lactate group

SUMMARY:
To assess the Influence of early lactate clearance rate monitoring in patients with sepsis.

ELIGIBILITY:
Inclusion Criteria:

* All patients whose blood lactate level reached or exceeded 2.0 mEq / L

Exclusion Criteria:

* Incomplete clinical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe sepsis or septic shock were recruited from Emergency ICU of the second hospital of Hebei Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-02-15 (Estimated)

PRIMARY OUTCOMES:
In-hospital 60days mortality | In-hospital 60 days
  In-hospital up to 60 days mortality of sepsis
ICU mortality | up to 30 days
  ICU up to 30 days mortality of sepsis

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No